CLINICAL TRIAL: NCT07344870
Title: Impact of Short-Term Parental Nutrition Education on the Performance and Body Composition of Young Basketball Players: A Pre-Post Intervention Study
Brief Title: Parental Nutrition Education on the Performance and Body Composition of Young Basketball Players
Acronym: PNE-YBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Mustafa Ozgur, Assistant Professor, Burdur Mehmet Akif Ersoy University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GO 2023/206; 1919B012306151 (Other Grant/Funding Number: TÜBİTAK the 2209-A University Students Research Projects Support Program)
Record Dates: First submitted 2025-12-09; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Nutritional Status; Athletic Performance; Body Composition; Adolescent; Healthy Diet
Keywords: Young players; physical performance; anthropometric measurement; nutrition education; parental involvement; dietary assessment

STUDY DESIGN:
Intervention Model Description: All participants were assigned to a single intervention arm receiving the parental nutrition education program. Efficacy was evaluated by comparing baseline (pre-intervention) measurements with post-intervention measurements (4 weeks later) within the same subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parental Nutrition Education Group (Experimental): Participants in this arm are young basketball players whose parents received a structured 4-week nutrition education program. The intervention included weekly 45-minute face-to-face seminars and printed educational materials covering macronutrients, hydration, and meal timing.
  Interventions: Behavioral: Parental Nutrition Education Program

INTERVENTIONS:
Behavioral: Parental Nutrition Education Program — All participants were assigned to a single intervention arm receiving the parental nutrition education program. Efficacy was evaluated by comparing baseline (pre-intervention) measurements with post-intervention measurements (4 weeks later) within the same subjects.

SUMMARY:
This study investigates the impact of a structured, short-term parental nutrition education program on the body composition, athletic performance, and dietary habits of young basketball players aged 8-13 years. Adolescence represents a critical window for physical growth and athletic development, yet many young athletes fail to meet nutritional recommendations. Given that parents are the primary food providers and decision-makers for children in this age group, their nutritional literacy is hypothesized to directly influence the athlete's diet and physical development.

The intervention consists of a 4-week nutrition education program provided to parents. The study utilizes a single-group pre-post design to evaluate changes in the athletes' Lean Body Mass (LBM), body fat percentage, athletic performance (encompassing vertical jump, sprint speed, and flexibility), and daily macronutrient intake (protein and carbohydrate) from baseline to post-intervention.

DETAILED DESCRIPTION:
Study Design: This study employs a single-group, pre-post quasi-experimental design to evaluate the efficacy of a parental nutrition education program. The study population consists of young basketball players aged 8-13 years recruited from the Burdur Mehmet Akif Ersoy University youth basketball team.

Intervention: The primary intervention is a structured "Parental Nutrition Education Program." The education is delivered to the parents/legal guardians of the athletes, as they are the primary food providers. The intervention consists of:

A comprehensive 90-minute online seminar (via Zoom) conducted by a registered dietitian. Topics include macronutrients (carbohydrates, proteins, fats), micronutrients (calcium, iron, vitamins), hydration strategies, meal timing (pre- and post-training nutrition), and healthy food choices .

Distribution of printed educational brochures and guides to reinforce the seminar content.

Q&A sessions to address specific nutritional concerns. The intervention period lasts for 4 weeks.

Data Collection and Procedures: Assessments are conducted at two time points: Baseline (Week 0) and Post-Intervention (Week 4).

Dietary Assessment: Dietary intake is evaluated using 3-day food consumption records (2 weekdays and 1 weekend day) via the retrospective recall method. Data are analyzed using the Nutrition Information System (BEBIS 8.0) to calculate daily energy, macronutrient, and micronutrient intake.

Anthropometric Measurements:

Body weight and height are measured using standard protocols. - Body composition (lean body mass, body fat percentage, and basal metabolic rate) is assessed using a bioelectrical impedance analysis (BIA) device (Tanita MC-780) under standardized conditions (fasted state, no exercise 12h prior).

Waist and hip circumferences are measured using a non-elastic tape. Performance Testing: Physical performance is assessed using a battery of field tests: - Speed: 20-meter sprint test using photocell timing gates. - Explosive Power: Vertical jump test using the Smart Jump System and Standing Long Jump test. - Strength: Handgrip strength (right and left) using a digital dynamometer (Takei 5401). - Endurance: Maximum number of push-ups and sit-ups in 30 seconds. - Agility: T-test. - Flexibility: Sit-and-reach test.

Nutrition Knowledge: The sports nutrition knowledge level of parents is assessed using the "Sports Nutrition Knowledge Level Test" (SNKT), adapted into Turkish, consisting of 20 questions.

Statistical Analysis: Pre- and post-intervention data are compared using paired sample t-tests (for normally distributed data) or Wilcoxon signed-rank tests (for non-normal data). A responder analysis is conducted by stratifying participants based on the change in their protein intake to evaluate dose-response relationships.

ELIGIBILITY:
Inclusion Criteria:

* Boy and girl basketball players aged 8 to 13 years.
* The youth basketball team must include active licensed players.
* The candidate must maintain regular attendance at training sessions (at least 3 days per week).
* Parents must be willing to participate in the education program and provide written informed consent.

Exclusion Criteria:

* Diagnosed with chronic metabolic or hormonal diseases.
* Musculoskeletal injuries within the last 3 months.
* Use of medications or supplements affecting metabolism.
* Failure to maintain regular training attendance.
* Parents withdrawing consent during the study.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Lean Body Mass | Baseline (Week 0) and Post-intervention (Week 4).
  Body composition was assessed using a Bioelectrical Impedance Analysis (BIA) device (Tanita MC-780) under standardized fasting conditions. The outcome measures the change in lean body mass (kg) from baseline to the end of the intervention

SECONDARY OUTCOMES:
Change in Athletic Performance Parameters | Baseline (Week 0) and post-intervention (Week 4).
  Performance was evaluated using a battery of field tests: Flexibility (cm), Reaction (cm), Vertical jump (cm), Standing long jump (cm)
Change in Athletic Performance Parameters-2 | Baseline (Week 0) and Post-intervention (Week 4)
  Right and Left Hand-claw strength (kg)
Change in Athletic Performance Parameters-3 | Baseline (Week 0) and Post-intervention (Week 4)
  Count of repetitions The maximum number of push-ups and sit-ups that can be completed within a set time.
Change in Daily Dietary Intake-1 | Baseline (Week 0) and post-intervention (Week 4).
  The assessment was conducted using 3-day food consumption records, using the retrospective recall method. Daily intake of energy kcal/day
Change in Daily Dietary Intake-2 | Baseline (Week 0) and post-intervention (Week 4).
  The assessment was conducted using 3-day food consumption records, using the retrospective recall method. Daily intake of macronutrients (carbohydrate, protein, and fat) (g/day)
Change in Daily Dietary Intake-3 | Baseline (Week 0) and post-intervention (Week 4).
  The assessment was conducted using 3-day food consumption records, using the retrospective recall method. Daily intake of micronutrients (mcg/day) was analyzed using the Nutrition Information System (BEBIS).

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available upon reasonable request to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Result] American College of Sports Medicine. ACSM's Guidelines for Exercise Testing and Prescription. 8th ed. Philadelphia, PA: Lippincott Williams & Wilkins; 2002
- [Result] Keser A, Binnetoğlu FK, Asil E, Babaoglu K. Comparison of food consumption and nutritional statuses of athletic adolescents. Anthropologist. 2016;25(1-2):60-69. doi:10.1080/09720073.2016.11892089
- [Result] Dener B. Voleybol oyuncularının beslenme bilgi düzeyi ile beslenme durumunun değerlendirilmesi ve beslenme eğitiminin etkisi [master's thesis]. Ankara: Sağlık Bilimleri Enstitüsü; 2018
- [Result] Torres-McGehee TM, Pritchett KL, Zippel D, Minton DM, Cellamare A, Sibilia M. Sports nutrition knowledge among collegiate athletes, coaches, athletic trainers, and strength and conditioning specialists. J Athl Train. 2012 Mar-Apr;47(2):205-11. doi: 10.4085/1062-6050-47.2.205. PMID 22488287

DOCUMENTS (1):
  • Study Protocol (2025-12-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT07344870/Prot_000.pdf